CLINICAL TRIAL: NCT05315024
Title: Prevalence, Genetic Risk Factor and the Use of Intradermally-administered Inactivated Influenza Vaccine With Topical Imiquimod in Influenza Vaccine Non-responsive Children
Brief Title: Influenza Vaccine With Topical Imiquimod in Influenza Vaccine Non-responsive Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Gilbert Chua, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-290
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repeat 0.5ml IM Quadrivalent IIV (IIV-IM) (Experimental): Repeat 0.5ml IM Quadrivalent IIV (IIV-IM) (15micrograms haemagglutinin per vaccine strain)
  Interventions: Drug: Fluarix Tetra
- 0.1ml ID Quadrivalent IIV (IIV-ID) (Experimental): 0.1ml ID Quadrivalent IIV (IIV-ID) (3micrograms haemagglutinin per vaccine strain)
  Interventions: Drug: Fluarix Tetra
- 0.1ml ID Quadrivalent IIV (Experimental): 0.1ml ID Quadrivalent IIV (3micrograms haemagglutinin antigen per vaccine strain) + 5% imiquimod cream (IIV-Q-ID)
  Interventions: Drug: Fluarix Tetra; Drug: Imiquimod cream

INTERVENTIONS:
Drug: Fluarix Tetra — Fluarix Tetra
Drug: Imiquimod cream — Imiquimod cream
  Arms: 0.1ml ID Quadrivalent IIV

SUMMARY:
Aims and hypotheses to be tested:

Primary objective

- To compare the IIV responses, in terms of seroconversion rates, using ID IIV with topical 5% imiquimod (IIV-Q-ID), ID influenza vaccine alone (IIV-ID), and the second dose of IM influenza vaccine (IIV-IM) among children who are IIV non-responders.

Secondary objectives

* To determine the IIV non-responder rate in healthy Hong Kong children.
* To investigate the association between HLA molecules and IIV non-responsiveness.

Hypotheses

* The investigators hypothesize that among IIV non-responder children, the seroconversion rate after ID IIV with topical imiquimod will be significantly higher than a second IM IIV dose.
* The investigators hypothesize that the IIV non-responder rate is approximately 5-10% in the paediatric population.
* The investigators hypothesize that certain HLA alleles are associated with IIV non-responders.

DETAILED DESCRIPTION:
This study is a cross-over randomized-controlled trial (RCT). The outline of the study is shown in Figure 1. This study is divided into two parts: (i) screening for vaccine non-responders; and (ii) RCT for vaccine responsiveness using second dose IIV-IM, IIV-ID or IIV-Q-ID.

Children and adolescents between 8 and 18 years old will be recruited through our network of primary and secondary schools that have participated the Seasonal Influenza Vaccination School Outreach Programme before the influenza vaccination campaign. Information sheets, a consent form and a health demographics form indicating that they fulfill the inclusion and exclusion criteria (see below) will be distributed to the parents through the participating schools. A study hotline will be available for parents to contact the study team to answer any enquiries.

In the health demographics form, apart from questions related to the inclusion and exclusion criteria, the study team will also enquire about the subjects' demographics, including birth, gender, past medical history, and body weight and height. Previous influenza vaccination history will also be sought, including age at receiving the first influenza vaccine, whether the subjects have received influenza vaccines in the last season and the type of influenza vaccines they received.

All subjects should be receiving 0.5ml IM quadrivalent IIV, which contains 15micrograms hemagglutinin of each influenza strain, through the Seasonal Influenza Vaccination School Outreach Programme. Consented subjects will have 5-10ml clotted blood and 3ml EDTA blood draw at day 21 post-vaccination at school by our outreach study team. The parents of all participating subjects will receive an incentive equivalent to HKD 100. They will also receive their influenza vaccine response results in concealed envelops distributed through the schools.

Post-vaccination HAI titer against the Influenza B Yamagata strain ≤10 will be considered as "preliminary no seroconversion". The same serum taken on day 21 post-vaccination will be further processed to confirm that their HAI titer against the other Influenza A H1N1 and H3N2 and Influenza B Victoria strains are also ≤10. MN assay for all four strains will also be performed as the baseline for the part 2 RCT.

Non-responders will be called back to attend a research clinic and will be randomized to one of the following revaccination strategies: (i) repeat 0.5ml IM Quadrivalent IIV (IIV-IM) (15micrograms haemagglutinin per vaccine strain); (ii) 0.1ml ID Quadrivalent IIV (IIV-ID) (3micrograms haemagglutinin per vaccine strain); or (iii) 0.1ml ID Quadrivalent IIV (3micrograms haemagglutinin antigen per vaccine strain) + 5% imiquimod cream (IIV-Q-ID). Subjects randomized to receive 5% imiquimod cream will have the injection site disinfected by 70% alcohol swab followed by application of the imiquimod cream for 5 minutes before the intradermal injection over a 16cm2 skin area of the deltoid described in previous studies. 0.1ml IIV, which contains 3micrograms hemagglutinin of each influenza strain, will be administered intradermally using a MicronJetTM microneedle. All subjects will be observed for 15 to 30 minutes in the waiting area for any local adverse reactions. These subjects will be called back on day 7 and 21 after the second dose of vaccination for blood testing. 5- 10ml clotted blood will be obtained to measure the vaccine response. HAI and MN assays against the four vaccine strains will be performed.

To determine the association between HLA alleles and IIV non-responsiveness, HLA genotyping will be performed among non-responders and responders in 1:2 ratios. Assuming that there will be 72-100 IIV non-responders from our cohort, HLA genotyping will be performed in 200 age- and gender-matched IIV responder controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years old
* Subjects receiving IIV influenza vaccination through the Seasonal Influenza Vaccination School Outreach Programme.

Exclusion Criteria:

* Age <8 years old to avoid the need for second dose vaccine in case the subjects have never had influenza vaccines before
* Age >18 years old
* Received any forms of influenza vaccines, including the intranasal live-attenuated influenza vaccines or inactivated vaccines, in the past six months
* Underlying chronic illnesses, including immunodeficiencies or autoimmune diseases
* Using immunosuppressive reagents, such as long-term corticosteroids, and other steroid-sparing reagents 6 months prior to the recruitment
* Received intravenous immunoglobulin or other blood products 3 months prior to the recruitment
* Had upper respiratory tract infection symptoms within two weeks before the vaccination, including fever, cough, sore throat, and coryza
* Previous allergic reactions to imiquimod, influenza vaccines, and their excipients.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The IIV responses, in terms of seroconversion rates, using ID IIV with topical 5% imiquimod (IIV-Q-ID), ID influenza vaccine alone (IIV-ID), and the second dose of IM influenza vaccine (IIV-IM) among children who are IIV non-responders | 2 years

SECONDARY OUTCOMES:
The IIV non-responder rate in healthy Hong Kong children. The association between HLA molecules and IIV non-responsiveness. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert T Chua, Principal Investigator — The University of Hong Kong